CLINICAL TRIAL: NCT04578184
Title: Comparison of Two Optical Coherence Tomography Devices in Corneal Epithelial Thickness Maps
Brief Title: Epithelial Thickness Map
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of Department of Ophthalmology, Professor, Principal Investigator, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Epithelial thickness map
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epithelial thickness map evaluation in keratoconus patients (Other): Patients included in the study will be measured with the corneal acquisition mode, also allowing for epithelium thickness data, on each device without pupil dilatation Each patient will be measured three times with both devices. The corneal epithelial thickness will be measured as the distance between the air-tear and the epithelium-Bowman interfaces.
  Interventions: Diagnostic Test: Corneal epithelial thickness measurements
- Epithelial thickness map evaluation in healthy cornea patients (Other): Patients included in the study will be measured with the corneal acquisition mode, also allowing for epithelium thickness data, on each device without pupil dilatation Each patient will be measured three times with both devices. The corneal epithelial thickness will be measured as the distance between the air-tear and the epithelium-Bowman interfaces.
  Interventions: Diagnostic Test: Corneal epithelial thickness measurements

INTERVENTIONS:
Diagnostic Test: Corneal epithelial thickness measurements — Corneal epithelial thickness measurements using two optical coherence tomography devices in healthy and keratoconus corneas.

SUMMARY:
In keratoconic eyes, the corneal epithelium shows a localized thinning over the cone that is surrounded by an annulus of epithelial thickening. It has been postulated that epithelial thickness mapping can be a sensitive tool for the keratoconus diagnosis. In keratoconus screening the 5 mm diameter of the corneal centrum may be sufficient while studies have shown that the cone apex is located in this area.

Aim of this study is to assess agreement and repeatability of epithelial thickness measurements using two optical coherence tomography devices in healthy and keratoconus corneas.

Secondary objective is to evaluate the differences between healthy and keratoconus eyes using epithelial thickness map data.

This is a prospective monocentric study that includes patients divided into two groups: patients with keratoconus and a control group formed out of patients without corneal pathologies. For each patient only one eye will be included and corneal measurements will be performed, focused on the corneal epithelium thickness.

DETAILED DESCRIPTION:
In total 50 eyes of 50 patients will be included, divided into two groups: study group comprised of 20 eyes with diagnosed keratoconus and a control group formed out of 30 healthy eyes.

Patients included in the study will be measured with the corneal acquisition mode, also allowing for epithelium thickness data, on each device without pupil dilatation. After each measurement patients will be asked to blink in order to allow adequate tear-film recovery. Each patient will be measured three times with both devices. Only one visit will be necessary.

The order in which the measurements will be performed (Anterion or MS-39) will be randomised using randomised.org.

The corneal epithelial thickness will be measured as the distance between the air-tear and the epithelium-Bowman interfaces.

Main outcome variable:

- Mean differences in central corneal epithelial thickness between the devices investigated (+ limits of agreement (1.96xSD) between the investigated devices)

Secondary outcome variables:

* Repeatability coefficient (within subject standard deviation - SD) and coefficient of variation of the two devices
* Comparison in epithelial thickness between normal and keratoconus eyes
* Sensitivity and specificity of swept-source OCT device in keratoconus diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosed keratoconus (diagnosed using tomography and topography map changes and slit-lamp changes) and patients with healthy cornea
* Age 21 and older
* Signed informed consent

Exclusion Criteria:

* Previous ocular surgery
* Associated corneal pathologies (e.g. trauma, edema, scarring)
* In women of childbearing age, a pregnancy test will be performed before inclusion into the study.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Agreement between two ss-OCT devices in corneal epithelial thickness measurements (LoA in micrometer) | 6 months

SECONDARY OUTCOMES:
Repeatability between two ss-OCT devices in corneal epithelial thickness measurements (determination of within-subject standard deviation and Coefficient of variation) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof., MD, Principal Investigator — Head of Department of Ophthalmology, Professor, Principal Investigator
Locations (1):
- Hanusch Hospital, Ophthalmology Department, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No